CLINICAL TRIAL: NCT03563365
Title: A Randomized, Investigator Blinded, Single Site, Three Arm Clinical Study to Assess the Functional and Emotional Benefits of Replenix Power of Three Cream With Resveratrol , Replenix Power of Three Cream With Resveratrol With Adapalene and Benzoyl Peroxide Gel, 0.1%/2.5%, and Adapalene and Benzoyl Peroxide Gel, 0.1%/2.5%, Utilized to Treat Subjects With Facial Acne Vulgaris
Brief Title: The Functional and Emotional Benefits of Replenix Power of Three With Resveratrol
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Yardley Dermatology Associates (Other)
Collaborators: Topix Pharmaceuticals, Inc (Unknown)
Responsible Party: Principal Investigator, Michelle Sibona, Principal Investigator/ Clinical Director, Yardley Dermatology Associates
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TPX-PW3-2018-A
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Resveratrol; Adapalene

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Subject is instructed not to discuss or disclose treatment arm with PI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Replenix (Experimental): Replenix power of 3 cream with Resveratrol applied twice daily
  Interventions: Other: Replenix Power of 3 Cream with resveratrol
- Replenix and Adapalene and Benzoyl Peroxide gel (Experimental): Replenix power of 3 cream with Resveratrol applied twice daily and Adapalene and Benzoyl Peroxide Gel, 0.1%/2.5% applied once daily
  Interventions: Other: Replenix Power of 3 Cream with resveratrol; Drug: Adapalene and Benzoyl peroxide gel, 0.1%/2.5%
- Adapalene and Benzoyl Peroxide gel (Active Comparator): Adapalene and Benzoyl Peroxide Gel, 0.1%/2.5% applied once daily
  Interventions: Drug: Adapalene and Benzoyl peroxide gel, 0.1%/2.5%

INTERVENTIONS:
Other: Replenix Power of 3 Cream with resveratrol — Cosmetic product containing Green Tea Polyphenols, Resveratrol, Caffeine USP, Bisabolol Cucumber extract, Chamomile extract, Rosemary extract, Squalane, Soy Phospholipids
  Arms: Replenix; Replenix and Adapalene and Benzoyl Peroxide gel
Drug: Adapalene and Benzoyl peroxide gel, 0.1%/2.5% — FDA approved topical agent for the treatment of acne
  Arms: Adapalene and Benzoyl Peroxide gel; Replenix and Adapalene and Benzoyl Peroxide gel

SUMMARY:
A Randomized, Investigator Blinded, Single Site, Three Arm Clinical Study to Assess the Functional and Emotional Benefits of Replenix Power of Three Cream with Resveratrol , Replenix Power of Three Cream with Resveratrol with Adapalene and Benzoyl Peroxide Gel, 0.1%/2.5%, and Adapalene and Benzoyl Peroxide Gel, 0.1%/2.5%, utilized to treat subjects with Facial Acne Vulgaris

DETAILED DESCRIPTION:
Acne vulgaris is a common skin problem which can be challenging to treat. Enhancing the efficacy and tolerability of treatment regimens can enhance compliance and outcomes thereby potentially decreasing the morbidities associated with acne vulgaris.

The present study is designed to assess the ability of Power of 3 with resveratrol to improve efficacy and tolerability of an existing combination acne medication.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of Acne vulgaris
2. On the face, ≥ 20 non-inflammatory lesions (i.e., open and closed comedones) AND < 75 inflammatory lesions (i.e., papules and pustules) AND ≤ 1 nodulocystic lesions (i.e., nodules and cysts).
3. Investigator's Global Assessment (IGA) of acne severity grade 2 or 3
4. Subject must be able to follow study instructions and likely to complete all required visits, as assessed by the Investigator.
5. Subject/Guardian must sign an IRB-approved Informed Consent/Assent/Assent Form including photography consent, and the Authorization for Use and release of Health and Research Study Information (HIPAA) form prior to any study-related procedures being performed

Exclusion Criteria:

1. Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).
2. Subjects who have acne conglobata, acne fulminans and secondary acne (e.g.:

   chloracne and drug induced acne).
3. Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris. Well trimmed moustaches are allowed.
4. History of hypersensitivity or allergy to benzoyl peroxide or adapalene and or any of the study product ingredients.
5. Subjects who have a severe or intense irritation on the face.
6. Use within 6 months prior to baseline (Randomization) of oral retinoids (e.g. Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
7. Use for less than 3 months prior to baseline (Randomization) of estrogens or oral contraceptives; use of such therapy is allowed if it will remain constant throughout the study.
8. Use on the face within 1 month prior to baseline (Randomization) or during the study of: 1) cryodestruction or chemodestruction, 2) dermabrasion, 3) photodynamic therapy, 4) acne surgery, 5) intralesional steroids, or 6) x-ray therapy.
9. Use within 1 month prior to baseline (Randomization) of: 1) spironolactone, 2) systemic steroids, 3) systemic antibiotics, 4) systemic treatment for acne vulgaris (other than oralretinoids, which require a 6-month washout), or 5) systemic anti- inflammatory agents.
10. Use within 2 weeks prior to baseline (Randomization) of: 1) topical steroids, 2) topical retinoids, 3) topical acne treatments including over-the-counter preparations, 4) topical anti-inflammatory agents, 5) medicated cleansers or 6) topical antibiotics.
11. Subjects who have had general anesthesia for any reason and patients who have received neuromuscular blocking agents within 14 days prior to study entry (Randomization).
12. Concomitant use of facial product containing glycolic or other acids, masks, washes or soaps containing benzoyl peroxide or salicylic acid, non mild cleansers or moisturizers containing retinol, salicylic or α- or β-hydroxy acids.
13. Concomitant use of mega-doses of certain vitamins (such as vitamin D and vitamin B12), haloperidol, halogens such as iodide and bromide, lithium, hydantoin and phenobarbital.
14. Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the past 2 weeks or during the study.
15. Concomitant use of tanning booths or sunbathing.
16. A significant medical history of or are currently immunocompromised
17. Have any systemic or dermatologic disease that may affect the evaluation of study results.
18. Have a history of regional enteritis, ulcerative colitis, pseudomembranous colitis or antibiotic-associated colitis.
19. Subjects with clinically significant unstable medical disorders, life-threatening disease, or current malignancies.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment (IGA) | Screening, Baseline, Week 2, Week 4, Week 8, Week 12
  To assess the change in Acne Vulgaris on a scale of 1 to 4, where 1 represents clear skin and 4 represents severe acne, at each scheduled visit with the use of Replenix Power of three with Resveratrol.
Subject Global Assessment (SGA) | Screening, Baseline, Week 2, Week 4, Week 8, Week 12
  To assess the change in Acne Vulgaris on a scale of 1 to 5, where 1 represents a worsening of acne and 5 represents clearing of acne, at each scheduled visit as compared to baseline with the use of Replenix Power of three with Resveratrol.
Subject Overall Assessment of Tone and Texture (SOATT) | Screening, Baseline, Week 2, Week 4, Week 8, Week 12
  To assess the change on skin tone and texture on a scale of 1 to 7, where 1 represents worse tone and texture and 7 represents better tone and texture, at each scheduled visit with use of Replenix Power of three with Resveratrol.
Investigator Overall Assessment of Tone and Texture (IOATT) | Screening, Baseline, Week 2, Week 4, Week 8, Week 12
  To assess the change on skin tone and texture on a scale of 1 to 7, where 1 represents worse tone and texture and 7 represents better tone and texture, at each scheduled visit with use of Replenix Power of three with Resveratrol.
Subject Assessment of Skin Dysesthesia (SDA) | Screening, Baseline, Week 2, Week 4, Week 8, Week 12
  To assess the change in Dysesthesia on a scale of 1 to 7, where 1 represents no dysesthesia and 7 represents severe dysesthesia, at each scheduled visit with use of Replenix Power of three with Resveratrol.
Subject Quality of Life (SQOL) | Screening, Baseline, Week 12
  To assess the change in Subject Quality of Life on a scale of 1 to 7, where 1 represents better quality of life and 7 represents worse quality of life, at Screening, Baseline and week 12 with use of Replenix Power of three with Resveratrol.
Local Tolerability Assessment | Screening, Baseline, Week 2, Week 4, Week 8, Week 12
  To assess the change in Local Tolerability on a scale of 0 to 3, where 0 represents no tolerability issues and 3 represents severe tolerability issues, at each scheduled visit with use of Replenix Power of three with Resveratrol.

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Fried, MD, PhD, Principal Investigator — Yardley Dermatology Associates, PC
Locations (1):
- Yardley Dermatology Associates, PC, Yardley, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No